CLINICAL TRIAL: NCT04477018
Title: 16 Weeks' Dietary Supplementation With Iron and Iron + Vitamin C on Cerebral Blood Flow and Energy Expenditure in Women of Reproductive Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 9BN2
Record Dates: First submitted 2020-07-09; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Iron; Cerebral Blood Flow; Energy Metabolism; Cognitive Function
Keywords: Iron supplementation; Cerebral blood flow; Near infrared spectroscopy; Indirect calorimetry; Energy metabolism
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Participants will receive either iron and vitamin C, iron alone or placebo for a period of 16 weeks to consume daily
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iron and Vitamin C (Experimental): 28 mg iron bis-glycinate chelate and 240 mg vitamin C
  Interventions: Dietary Supplement: Iron bis-glycinate chelate and vitamin C
- Iron (Active Comparator): 28 mg iron bis-glycinate chelate
  Interventions: Dietary Supplement: Iron bis-glycinate chelate
- Placebo (Placebo Comparator): Matched placebo tablets
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Iron bis-glycinate chelate and vitamin C — 28 mg iron; 240 mg vitamin C
  Arms: Iron and Vitamin C
Dietary Supplement: Iron bis-glycinate chelate — 28 mg iron only
  Arms: Iron
Dietary Supplement: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
Iron deficiency is the most prevalent nutritional deficiency worldwide with one in four estimated to be affected by iron deficiency anaemia. Women of reproductive age are at greatest risk for iron deficiency and anaemia due to iron losses during menstruation and childbirth as well as the increased need for iron throughout pregnancy. However, iron deficiency without anaemia is at least twice as common as iron deficiency anaemia with females aged 11-49 at the biggest risk of all. Despite this, it is commonly left undiagnosed. Those who are iron deficient non-anaemic can still suffer from the same common consequences of iron deficiency anaemia; these include unexplained fatigue, mood changes and decreased cognitive performance. It is postulated that for any cognitive and behavioural change to occur, a complementary change in neural functioning is required. A recent cross-sectional study has identified increases in cognitive demand to produce decrements in measures of cognitive performance and increases in brain activity and metabolic measures; the magnitude of such are evidenced to be directly related to iron status. However, such measures do not provide an estimate of overall oxygen consumption that is specific to the brain in order to be able to associate changes in cognitive performance and energy expenditure specifically to the brain itself. The current study aims to investigate the parallel effects of iron supplementation on cerebral haemodynamics and energy metabolism to determine the ability of iron to modulate whole body energy metabolism and utilisation of metabolic substrates at rest and during cognitive demand in a sample of non-anaemic iron deficient and iron sufficient women of reproductive age.

DETAILED DESCRIPTION:
Each participant will be required to attend the laboratory on four occasions. The first is comprised of a screening/training visit, which will take place in the afternoon for approximately 2.5 hours. This will also be between days 21-28/ the week before onset of their menstrual cycle. If they do not have menstrual bleeds then this appointment can be any afternoon. This will comprise: briefing of requirements of the study; obtaining of informed consent; confirmation of eligibility to take part, including collection of demographic data and health screening, and training on the cognitive and mood measures. The training session will follow standard operating procedures to decrease the chance of learning effects during main trials. Extra training will be given where necessary.

Participants will be required to complete questionnaires based upon food frequency, caffeine consumption and to estimate the number of hours of exercise completed on a weekly basis. A menstrual cycle questionnaire will also be completed to estimate menstrual blood loss and so that participants attend their testing visit during days 7-14 of their cycle. If participants do not have a menstrual cycle due to contraceptive methods, then appointments will be approximately two weeks apart. A finger-prick and venous blood sample will be collected from participants, which will be analysed for iron status. Those whose haemoglobin levels are <120g/L will be advised to seek advice from their GP. Participants who fell into the iron status category of iron sufficient (haemoglobin ≥120 g/L and serum ferritin > 20 µg/L) or non-anaemic iron deficient (haemoglobin ≥120 g/L and serum ferritin ≤ 20 µg/L) will be informed of their eligibility for the intervention study by email or phone between the initial visit and their next. This will include the option to enrol in an additional assessment of neuroimaging and energy metabolism.

For the testing visit, participants will be asked to fast for 12 hours prior to the visit, avoiding intake of all food and drink with the exception of water. They will also be asked to avoid alcohol and refrain from intake of 'over the counter' medication for 24 hours. Participants will arrive at the laboratory at a designated time in the morning. The following procedures will take place prior to cognitive and mood testing:

Review of continued conformity to eligibility criteria Adverse event and concomitant medication assessment Ensure that participant is in good health

Participants will then complete the baseline cognitive and mood assessments. Following this, participants are informed of their iron status and will be briefed regarding the requirements of the intervention study and additional assessment. Following this, informed consent will be obtained prior to starting the additional assessment. Participants will have a frequency domain near-infrared spectroscopy headband attached to the forehead to measure cerebral blood flow at rest for five minutes. Following this, participants will instead have a continuous wave near-infrared spectroscopy headband attached to the forehead to measure cerebral blood flow, and a face mask fitted to measure expired air. Participants will have another five minute rest before completing an additional battery of cognitive tasks for approximately 35-40 minutes. Once complete, participants will be randomised to one of three treatments and be provided with a treatment diary to log treatment consumption and any adverse events experienced.

Participants will return to the laboratory after 8 weeks to exchange treatment bottles and diaries in order to check compliance.

Participants will finally return to the laboratory after a further 8 weeks (16 weeks total). The same procedures will take place prior to cognitive and mood testing as completed at the baseline testing visit, with the addition of finger prick and venous blood sample and weight measurement. Participants will then complete the same cognitive, mood and neuroimaging and energy metabolism assessments as completed during the baseline testing visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Female
* Aged 18-49 (inclusive)
* Have a BMI of between 18.5-40
* Have an English bank account (required for payment)

Exclusion Criteria:

* Aged under 18 or above 49 years
* BMI lower than 18.5 or higher than 40
* Pre-existing medical condition/illness with some exceptions - please check with researcher
* Blood disorders (including anaemia) or any known active infections
* Current or past breast cancer diagnosis and/or mastectomy
* Smoking or use of any nicotine replacement products e.g. vaping, gum, patches
* Pregnant, trying to get pregnant or breast feeding
* Currently taking any prescription medication with some exceptions - please check with researcher
* Food allergies/sensitivities relevant to the study
* Regular use of dietary/herbal supplements within the last month (defined as more than 3 consecutive days or 4 days in total)
* Use of iron supplements within the past 4 months
* Have donated more than 300ml of blood in the past 3 months
* Have haemoglobin levels below 120g/L
* History of significant head trauma or suffer from frequent migraines that require medication (more than or equal to one per month)
* Learning difficulties, dyslexia, or colour blindness
* Visual impairment that cannot be corrected with glasses or contact lenses
* Currently taking part in any other clinical or nutritional intervention studies or have in the past 4 weeks
* Any health condition that would prevent fulfilment of the study requirements

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must be female at birth
Enrollment: 78 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-06-08 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow | 16 weeks
  Near Infrared Spectroscopy outcomes for cerebral blood flow measurement at rest and during cognitive demand

SECONDARY OUTCOMES:
Serial Subtraction Performance | 16 weeks
  Performance on serial subtractions (3s and 7s) will be assessed as total responses and total errors
Rapid Visual Information Processing | 16 weeks
  Performance is assessed as accuracy (%), correct reaction time (msec) and false alarms
Subjective alertness | 16 weeks
  Subjective alertness will be derived from an Alertness visual analogue scale presented following cognitive task performance. Scores range from 0 to 100. Higher scores are indicative of greater feelings of alertness.
Subjective fatigue | 16 weeks
  Subjective mental fatigue will be derived from a Mental Fatigue visual analogue scale presented following cognitive task performance. Scores range from 0 to 100. Higher scores are indicative of greater feelings of mental fatigue.
Fat Oxidation | 16 weeks
  Fat oxidation will be assessed through indirect calorimetry at rest and during cognitive demand
Carbohydrate Oxidation | 16 weeks
  Carbohydrate oxidation will be assessed through indirect calorimetry at rest and during cognitive demand
Respiratory Energy Ratio | 16 weeks
  Respiratory energy ration will be assessed through indirect calorimetry at rest and during cognitive demand
Total Energy Expenditure | 16 weeks
  Total energy expenditure will be assessed through indirect calorimetry at rest and during cognitive demand

CONTACTS AND LOCATIONS:
Locations (1):
- Brain, Performance & Nutrition Research Centre, Northumbria University, Newcastle upon Tyne, United Kingdom